CLINICAL TRIAL: NCT01840774
Title: Modifying Virtual Reality Analgesia With Low-Dose Pain Medication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Sam Sharar, Study Principal Investigator, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 43929
Record Dates: First submitted 2013-04-08; First posted 2013-04-26 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Virtual Reality Therapy
MeSH Terms: interventions — Acetaminophen; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-dose pain medication (Active Comparator): 80min IV infusion of a low-dose pain medication
  Interventions: Drug: Low-dose pain medication (Ketalar) and saline placebo
- saline placebo (Placebo Comparator): 80min IV infusion of a saline placebo
  Interventions: Drug: Low-dose pain medication (Ketalar) and saline placebo

INTERVENTIONS:
Drug: Low-dose pain medication (Ketalar) and saline placebo

SUMMARY:
The purpose of this study is to determine how pain relief is modified when the investigators combine the Virtual Reality based Snow World game with certain pain medications.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, within subject 2x2 factorial, repeated measures study. Research participants will play two versions of the Virtual Reality based video game "Snow World" and be given thermal and electrical stimulus. Each of two study visits will be identical with the exception of whether or not the participant will receive an iv infusion of a low dose pain medication or a saline placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and females between the age of 18 and 60 years
* Ability to communicate orally
* Ability to read and understand English
* Body Mass Index between 20-35

Exclusion Criteria:

* Women who are pregnant, trying to become pregnant, or who are breastfeeding
* History of alcohol or substance abuse
* Major medical illness; including history of migraine headaches, seizures, brain injury, or peripheral neuropathy
* Current use of analgesics including acetaminophen, non-steroidal anti-inflammatories, or opioids
* Predisposition to severe motion sickness
* Unusual sensitivity or lack of sensitivity to pain
* Urine toxicology positive for opioids or benzodiazepines

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Pain responses between placebo and the low-dose pain medication while playing Snow World. We will assess pain responses with subjective questionnaires concerning the participant's experience while playing Snow World. | Conclusion of 120 study visits. Each participant will spend a total of 8 hours with us.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Sharar, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States